CLINICAL TRIAL: NCT06184256
Title: BfedBwell: Multiphase Optimization Strategy Pilot Trial of a Nutrition Intervention for Cancer Survivors With Overweight and Obesity
Brief Title: BfedBwell Optimization Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-2151.cc; 1K99CA287061-01 (NIH)
Record Dates: First submitted 2023-12-13; First posted 2023-12-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Survivorship; Cancer
Keywords: Overweight; Obesity; Diet, food, and nutrition; Exercise; Healthy lifestyle behaviors; Cancer
MeSH Terms: conditions — Neoplasms; Overweight; Obesity; Motor Activity | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Core Curriculum (Experimental): Participants will receive core curriculum
  Interventions: Behavioral: BfedBwell - Core Curriculum
- Core Curriculum and Group Support (Experimental): Participants will receive core curriculum and group support
  Interventions: Behavioral: BfedBwell - Core Curriculum; Behavioral: BfedBwell - Group Support
- Core Curriculum and Behavioral Skills (Experimental): Participants will receive core curriculum and behavioral skills
  Interventions: Behavioral: BfedBwell - Core Curriculum; Behavioral: BfedBwell - Behavioral Skills
- Core Curriculum, Behavioral Skills, and Group Support (Experimental): Participants will receive core curriculum, behavioral skills, and group support
  Interventions: Behavioral: BfedBwell - Core Curriculum; Behavioral: BfedBwell - Behavioral Skills; Behavioral: BfedBwell - Group Support
- Core Curriculum and 1:1 Counseling (Experimental): Participants will receive core curriculum and 1:1 counseling
  Interventions: Behavioral: BfedBwell - Core Curriculum; Behavioral: BfedBwell - 1:1 Counseling
- Core Curriculum,1:1 Counseling, and Group Support (Experimental): Participants will receive core curriculum, 1:1 counseling, and group support
  Interventions: Behavioral: BfedBwell - Core Curriculum; Behavioral: BfedBwell - 1:1 Counseling; Behavioral: BfedBwell - Group Support
- Core Curriculum, 1:1 Counseling, and Behavioral Skills (Experimental): Participants will receive core curriculum, 1:1 counseling, and behavioral skills
  Interventions: Behavioral: BfedBwell - Core Curriculum; Behavioral: BfedBwell - 1:1 Counseling; Behavioral: BfedBwell - Behavioral Skills
- Core Curriculum, 1:1 Counseling, Behavioral Skills, and Group Support (Experimental): Participants will receive core curriculum, 1:1 counseling, behavioral skills, and group support
  Interventions: Behavioral: BfedBwell - Core Curriculum; Behavioral: BfedBwell - 1:1 Counseling; Behavioral: BfedBwell - Behavioral Skills; Behavioral: BfedBwell - Group Support
- Program Provider (Experimental): Providers will deliver and evaluate one or more components of the diet or exercise interventions
  Interventions: Behavioral: Program delivery

INTERVENTIONS:
Behavioral: BfedBwell - Core Curriculum — 12-week core nutrition education curriculum + 12-week tapered maintenance curriculum
  Arms: Core Curriculum; Core Curriculum and 1:1 Counseling; Core Curriculum and Behavioral Skills; Core Curriculum and Group Support; Core Curriculum, 1:1 Counseling, Behavioral Skills, and Group Support; Core Curriculum, 1:1 Counseling, and Behavioral Skills; Core Curriculum, Behavioral Skills, and Group Support; Core Curriculum,1:1 Counseling, and Group Support
Behavioral: BfedBwell - 1:1 Counseling — Individual 1:1 counseling sessions with a registered dietitian
  Arms: Core Curriculum and 1:1 Counseling; Core Curriculum, 1:1 Counseling, Behavioral Skills, and Group Support; Core Curriculum, 1:1 Counseling, and Behavioral Skills; Core Curriculum,1:1 Counseling, and Group Support
Behavioral: BfedBwell - Behavioral Skills — Group-based behavioral skills development sessions
  Arms: Core Curriculum and Behavioral Skills; Core Curriculum, 1:1 Counseling, Behavioral Skills, and Group Support; Core Curriculum, 1:1 Counseling, and Behavioral Skills; Core Curriculum, Behavioral Skills, and Group Support
Behavioral: BfedBwell - Group Support — Structured group support sessions
  Arms: Core Curriculum and Group Support; Core Curriculum, 1:1 Counseling, Behavioral Skills, and Group Support; Core Curriculum, Behavioral Skills, and Group Support; Core Curriculum,1:1 Counseling, and Group Support
Behavioral: Program delivery — Delivery and evaluation of one or more intervention components
  Arms: Program Provider

SUMMARY:
Using the Multiphase Optimization Strategy (MOST) framework, an engineering-based approach to efficiently and systematically develop, optimize, and evaluate behavioral interventions, this study will test three components: (1) 1:1 counseling with a registered dietitian, (2) behavioral skills development, and (3) group support for delivery alongside a core nutrition curriculum within a clinical exercise oncology program.

DETAILED DESCRIPTION:
Individuals with experience in delivery of lifestyle (e.g., diet, physical activity) interventions will be recruited to deliver and evaluate the integrated BfedBwell intervention.

Cancer survivors with overweight/obesity who have completed active treatment will be recruited from the University of Colorado Anschutz Medical Campus for participation in a 6-month cluster-randomized 2^3-factorial pilot optimization trial of the BfedBwell intervention. Feasibility and acceptability will be evaluated. Exploration of intervention effect on adherence to cancer survivorship guidelines, body composition, and cardiometabolic indicators of health will be used to determine a set of components that demonstrate patterns of efficacy.

ELIGIBILITY:
Inclusion Criteria:

For program delivery staff:

1. Men and women
2. Age ≥ 18 years
3. Speak English
4. Self-reported previous experience in the delivery of nutrition, exercise, or behavioral weight management programs

For intervention participants:

1. Men and women
2. Age 18-75 years
3. BMI 25-45 kg/m2
4. History of cancer within the past 10 years with a diagnosis of an adulthood cancer of any type
5. In maintenance or surveillance status, defined as completion of active cancer therapy (e.g., surgery, radiation, chemotherapy, immunotherapy) with curative intent at least 3 months and no more than 10 years prior to enrollment or active surveillance with no treatment; ongoing targeted or hormone therapies ≥3 months prior to intervention start date and/or ongoing maintenance therapy ≥1 year is permitted (exceptions to this timeframe for completion of other therapies can be made on a case-by-case basis by the PI if patients are tolerating therapy without adverse effects and will have completed active treatment or been in stable maintenance treatment prior to the intervention start date)
6. Have a primary care provider (or are willing to establish care with a primary care provider prior to study enrollment) to address medical issues which may arise during screening or study procedures/interventions and who will provide clearance to participate in a nutrition and exercise program
7. Ability and willingness to participate in a supervised exercise program; with ability assessed by the Physical Activity Readiness Questionnaire (PAR-Q+) and questions based upon National Comprehensive Cancer Network (NCCN) guidelines (note: any positive responses will trigger a required physician clearance form)
8. Speak English
9. Have access to a computer or smart phone and Internet to join Zoom meetings, complete questionnaires, and access/download the True Coach virtual exercise coaching sessions
10. Live or work within 30 miles of the AHWC (exceptions may be made at the discretion of the study PI on a case-by-case basis for highly motivated subjects)
11. Not be planning for major elective surgery, to travel for >2 consecutive weeks, or relocate/move during the intervention (~6 months)
12. No nicotine or tobacco use within previous 6 months
13. Agree to refrain from use of all nutritional supplements aside from those prescribed by a physician for the duration of the study
14. Capable and willing to give informed consent and understand exclusion criteria
15. Willing to attend weekly small group education sessions and some, none, or all of the following: monthly behavioral skills development sessions, weekly group support sessions and/or monthly 1:1 counseling held by a registered dietitian (RD)
16. Willing to attend up to two BfitBwell exercise sessions (one in person, one virtual) per week for first 12 weeks then once monthly in person and once weekly virtual sessions for second 12 weeks
17. Not meeting dietary guidelines [i.e., Healthy Eating Index (HEI) score <80 as assessed via NCI DHQ III food frequency questionnaire] or physical activity guidelines [i.e., <150 minutes moderate/vigorous activity per week via self-report on Godin-Shephard Leisure-Time Physical Activity Questionnaire]

Exclusion Criteria

For program delivery staff:

None

For intervention participants:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status 2 or higher
2. Actively undergoing chemotherapy, radiation, immunotherapy with curative intent or within 3 months of completion of surgery, chemotherapy, or radiation treatment or recent initiation of targeted/hormonal therapy (<3 months) or maintenance therapy (<1 year) unless well-tolerated and deemed acceptable by PI on a case-by-case basis
3. Greater than 10 years post-active or maintenance therapy
4. Plans to relocate within the next 6 months
5. Plans for extended travel (>2 weeks) within the next 6 months
6. For females:

   1. Currently pregnant or lactating
   2. Pregnant within the past 6 months
   3. Planning to become pregnant in the next 18 months; sexually active women of childbearing potential may be enrolled if they have had a tubal ligation or use a reliable means of contraception
7. Any major surgery within the past 3 months or planned elective surgery during the intervention period, including mastectomy
8. Have completed treatment that significantly impacts digestion, metabolism, and/or food intake (e.g., surgical loss of esophagus, stomach, colon)
9. Recent (past 6 months) acute coronary event, unstable angina, coronary revascularization, stroke, or pulmonary embolism
10. Symptoms suggestive of cardiovascular disease (e.g., chest pain, shortness of breath at rest or with mild exertion, lightheadedness, syncope)
11. Uncontrolled hypertension, defined as diastolic blood pressure >100 mmHg, systolic blood pressure >160 mmHg, or resting heart rate >100 bpm as measured in duplicate on the screening visit after 5 minutes of rest in a seated position (if screening is needed due to lack of updated medical record within previous 12 months)
12. Diabetes (history of type 1 or type 2 diabetes, hemoglobin A1c ≥6.5%, or fasting glucose ≥126 mg/dL as measured during the screening visit if screening is needed due to lack of updated medical record within previous 12 months) unless well controlled on metformin or DPP-V inhibitor monotherapy with hemoglobin A1c <8%
13. History of uncontrolled thyroid disorder. History of thyroid disease or current thyroid disease treated with a stable medication regimen is acceptable
14. Triglycerides >500 mg/dL as measured on the screening visit (if screening is needed due to lack of updated medical record within previous 12 months)
15. LDL cholesterol >200 mg/dL as measured on the screening visit (if screening is needed due to lack of updated medical record within previous 12 months)
16. Presence or history of other metabolic or chronic health problems which would impact ability to safely participate in a weight loss intervention involving diet and exercise: significant cardiac arrhythmias or cardiac valvular disease, significant gastrointestinal, pulmonary, renal, musculoskeletal, neurologic, hematologic, or psychiatric disease
17. Have started lipid-lowering, hypertension, or oral hypoglycemic medication in previous 3 months
18. Sustained use of prescription or over-the-counter medications known to significantly impact appetite, weight, or energy metabolism (e.g., obesity pharmacotherapeutics agents, appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants) with the exception of anti-endocrine or Her2 directed treatment for breast cancer and standard of care anti-emetic or anti-diarrheal agents.
19. Sustained use of systemic glucocorticoids (current or in the past 6 months) unless physiologic replacement therapy for adrenal insufficiency
20. Previous obesity treatment with surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed >1 year before screening, (2) lap banding if the band has been removed >1 year before screening, (3) intragastric balloon if the balloon has been removed >1 year before screening, (4) duodenal-jejunal bypass sleeve if the sleeve has been removed >1 year before screening, or (5) AspireAssist or other endoscopically placed weight loss device if the device has been removed >1 year before screening
21. Participation within previous 6 months, current participation in, or planning to participate in any formal nutrition, weight loss, or physical activity programs or clinical trials over the next 6 months
22. Previous participation the BfitBwell exercise oncology program within the previous 3 years (exceptions may be made at the discretion of the study PI)
23. Nicotine or tobacco use (current or past 6 months)
24. Current alcohol or substance abuse as assessed by the Cut down, Annoyed, Guilty, and Eye-Opener (CAGE) questionnaire (note: study PI will follow up if screener raises any concerns of substance abuse to determine final eligibility)
25. History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder. Score >20 on the Eating Attitudes Test (EATS-26) or pattern of response on the Questionnaire of Eating and Weight Patterns (QEWP-5) suggestive of possible binge eating disorder or bulimia will require further assessment by the study MD to determine if it is appropriate for the subject to participate in the study
26. Current severe depression or history of severe depression within the previous year, based on Center for Epidemiologic Studies Depression Scale (CES-D) which in the opinion of the study MD would interfere with ability to adhere to the diet and exercise interventions and provide feedback on the interventions via questionnaires and focus groups
27. History of other significant psychiatric illness (e.g., psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the study MD would interfere with ability to adhere to the diet and exercise interventions and provide feedback on the interventions via questionnaires and focus groups
28. Have medical or physical limitations or contraindications to engaging in physical activity (e.g., severe orthopedic conditions, paralysis) or are considered high-risk based on ACSM guidelines
29. Are cognitively unable to consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Determine the research protocol recruitment feasibility of the BfedBwell nutrition intervention | 24 weeks
  Recruitment will be assessed as the number of adults screened and the proportion of eligible screens who enroll.
Determine the research protocol adherence feasibility of the BfedBwell nutrition intervention | 24 weeks
  Adherence will be assessed as [# sessions attended/# sessions provided] for each BfedBwell component.
Determine the research protocol outcome assessment feasibility of the BfedBwell nutrition intervention | 24 weeks
  Outcome assessment rates will be assessed as [# completing assessments/# enrolled].
Determine the research protocol retention feasibility of the BfedBwell nutrition intervention | 24 weeks
  Retention will be assessed as [# of participants who complete the 24-week intervention/# of participants randomized].
Determine the intervention acceptability by participants during focus groups | 24 weeks
  Participants will be asked to participate in a 90-minute focus group to provide qualitative feedback regarding their experience and satisfaction with the intervention.
Determine the intervention feasibility by program delivery staff using Feasibility of Intervention Measure (FIM) | 12 and 24 weeks
  Upon completion of the intervention, program delivery staff will be asked to complete the Feasibility of Intervention Measure (FIM). A Likert scale from 1 (completely disagree) to 5 (completely agree) is used for each question; higher scores indicate greater intervention feasibility.
Determine the intervention acceptability by program delivery staff using Acceptability of Intervention Measure (AIM) | 12 and 24 weeks
  Upon completion of the intervention, program delivery staff will be asked to complete the Acceptability of Intervention Measure (AIM). A Likert scale from 1 (completely disagree) to 5 (completely agree) is used for each question; higher scores indicate greater intervention acceptability.
Determine the intervention acceptability by program delivery staff using Intervention Appropriateness Measure (IAM) | 12 and 24 weeks
  Upon completion of the intervention, program delivery staff will be asked to complete the Intervention Appropriateness Measure (IAM). A Likert scale from 1 (completely disagree) to 5 (completely agree) is used for each question; higher scores indicate greater intervention appropriateness.
Determine the intervention acceptability by participants using the Net Promoter Score (NPS) | 12 and 24 weeks
  Participants will be asked to complete weekly ratings using the Net Promoter Score (NPS). Respondents are grouped as follows: 1) promoters (score 9-10) are loyal enthusiasts who will keep referring others and fueling growth, 2) passives (score 7-8) are satisfied but unenthusiastic customers who are vulnerable to competitive offerings, and 3) detractors (score 0-6) are unhappy customers who can impede growth with negative word-of-mouth. The final NPS score is calculated as % promoters - % detractors. NPS scores range from -100 to +100, with scores &gt;0 indicating good acceptability.

SECONDARY OUTCOMES:
Identify a set of components that demonstrate patterns of efficacy for increased adherence to lifestyle recommendations | 12 and 24 weeks
  Determine the change in adherence to cancer survivorship guidelines as measured by World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) scoring criteria. Scores range from 0 to 7 points. A higher score reflects greater adherence to the recommendations.
Identify a set of components that demonstrate patterns of efficacy for weight loss | 12 and 24 weeks
  Determine the change in weight as measured by digital scale. A lower weight indicates an improvement.
Identify a set of components that demonstrate patterns of efficacy for improvement in body composition | 12 and 24 weeks
  Determine the change in body composition as measured by dual x-ray absorptiometry (DXA). A lower body fat percentage indicates an improvement.
Measure the change in systolic blood pressure to determine improved cardiometabolic health | 12 and 24 weeks
  Systolic blood pressure will be measured at specific time points during the trial. A lower systolic blood pressure indicates an improvement.
Measure the change in diastolic blood pressure to determine improved cardiometabolic health | 12 and 24 weeks
  Diastolic blood pressure will be measured at specific time points during the trial. A lower diastolic blood pressure indicates an improvement.
Measure changes in total cholesterol to determine improved cardiometabolic health | 12 and 24 weeks
  Total cholesterol will be measured at specific time points during the trial. A lower total cholesterol indicates an improvement.
Measure changes in LDL cholesterol to determine improved cardiometabolic health | 12 and 24 weeks
  LDL cholesterol will be measured at specific time points during the trial. A lower LDL cholesterol indicates an improvement.
Measure changes in HDL cholesterol to determine improved cardiometabolic health | 12 and 24 weeks
  HDL cholesterol will be measured at specific time points during the trial. A higher HDL cholesterol indicates an improvement.
Measure changes in triglycerides to determine improved cardiometabolic health | 12 and 24 weeks
  Triglycerides will be measured at specific time points during the trial. Lower triglycerides indicate an improvement.
Measure changes in glucose to determine improved cardiometabolic health | 12 and 24 weeks
  Glucose levels will be measured at specific time points during the trial. Lower glucose levels indicate an improvement.
Measure changes in insulin to determine improved cardiometabolic health | 12 and 24 weeks
  Insulin levels will be measured at specific time points during the trial. Lower insulin levels indicate an improvement.
Intervention safety determined by number of adverse events | 12 and 24 weeks
  Overall rates of study-related mild, moderate, severe, and serious adverse events (AEs) will be tracked by study staff.

CONTACTS AND LOCATIONS:
Overall Officials: Emily B Hill, PhD, RDN, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States